CLINICAL TRIAL: NCT05047081
Title: Scoring Your College Goals: A Study to Increase Self-Efficacy in First-Year College Students
Brief Title: From Intention to Action:Scoring Your College Goals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Zucker Hillside Hospital (Other)
Collaborators: College of Staten Island, the City University of New York (Other)
Responsible Party: Principal Investigator, Timothy Michaels, PhD, Principal Investigator, The Zucker Hillside Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 21-0500
Record Dates: First submitted 2021-08-31; First posted 2021-09-16 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Depression; Anxiety
Keywords: Depression; Anxiety; College Mental Health; Mental Health Prevention
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- College Workshop Arm (Experimental): Intervention
  Interventions: Behavioral: Scoring Your College Goals Workshop
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Behavioral: Scoring Your College Goals Workshop — A two-hour virtual college readiness workshop.
  Arms: College Workshop Arm
Other: Placebo — Placebo Treatment-As-Usual Group which does not receive the workshop intervention
  Arms: Placebo

SUMMARY:
The current study aims to prevent the developmental of mental health symptoms in first-year college students through providing a workshop aimed at preparing students for the academic, social, and personal challenges associated with typical college experiences. Specifically, the study hypothesizes that first-year student students who participate in a workshop on college readiness will report fewer symptoms of depression and anxiety, higher levels of self-esteem, and better academic performance compared to a similar group of students who do not receive the intervention (the control group). Students in the intervention group will participate in a one-time, two-hour workshop that discusses expectations about college, setting goals that are aligned with one's values, predicting barriers to achieving these goals, and how to overcome these obstacles. The workshop will provide students with external resources (both on and off campus) for obtaining additional support to address barriers that arise during their college experiences. Students will complete questionnaires about symptoms of depression, anxiety, and their ability to cope with stress before the workshop, after the workshop, and at the end of their first semester. At the end of the Fall 2021 semester, students will be asked to share information about their Grade Point Average (GPA) and academic status. The investigators predict that at the end of the semester, those students who participated in the workshop will report lower levels of depression, anxiety and stress, higher levels of self-esteem, and a higher GPA compared to students who did not receive the intervention. Students who participated in the workshop will also be more likely to continue (enrolled in the Spring 2022 semester) compared to controls.

ELIGIBILITY:
Inclusion Criteria:

* First-year, first semester freshman enrolled in Psychology 100 courses at CUNY College of Staten Island.

Exclusion Criteria:

* Under 18 years old
* Violation of inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Self-Reported Depression Symptoms on the DASS-21 | Three Months
  Change in Depression Symptoms as measured by self-report on the Depression sub scale of the Depression, Anxiety and Stress Scale (DASS-21). Each sub scale of the DASS-21 has a range of 0-(lowest) to 42 (highest) with higher scores indicating worsening levels of psychopathology.
Change in Anxiety Symptoms as measured by the DASS-21 | Three Months
  Participants in the intervention arm but not the placebo group will demonstrate change in Depression Symptoms as measured by participant self-report on the Anxiety subscale of the Depression, Anxiety and Stress Scale (DASS-21).

SECONDARY OUTCOMES:
Change in self-efficacy as measured by the Coping Self-Efficacy Scale | Three Months
  Participants in the intervention group but not the control group will demonstrate significant change in self-reported self-efficacy scores as measured by the Coping Self-Efficacy Scale (CSE). Each sub scale of the CSE has a range of scores from 0 (lowest) to 60 (highest) with a higher score representing better (improved) coping self-efficacy.
Change in Coping abilities as measured by the Brief COPE | Three Months
  Participants in the intervention group but not the control group will demonstrate significant change in their ability to cope with stress as measured by self-reported total scores on the Brief COPE. The fourteen sub scales of the Brief COPE each have a range of 0 (lowest) to 8 (highest) with higher scores indicating higher levels of coping ability.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy I Michaels, PhD, Principal Investigator — The Zucker Hillside Hospital
Locations (1):
- CUNY College of State Island, Staten Island, New York, United States

IPD SHARING:
Plan to Share IPD: No